CLINICAL TRIAL: NCT03434834
Title: Advanced Angle-Resolved Low Coherence Interferometry (a/LCI) Systems for Improved Clinical Utility: An Optical Coherence Tomography (OCT) Pilot Study
Brief Title: OCT Pilot in Esophagus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00090173; R01CA210544 (NIH)
Record Dates: First submitted 2018-01-29; First posted 2018-02-15 (Actual); Results first posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-03

CONDITIONS: Barrett Esophagus
MeSH Terms: conditions — Barrett Esophagus | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- OCT of esophagus (Experimental): optical coherence tomography of esophagus
  Interventions: Device: optical coherence tomography

INTERVENTIONS:
Device: optical coherence tomography — OCT measurements of 5 locations in the esophagus

SUMMARY:
This is a pilot study to test a newly developed optical coherence tomography (OCT) device to determine 1) whether adequate tissue contact can be attained to acquire high quality images, and 2) to identify if these images can discern whether the imaged tissue is squamous or Barrett's Esophagus (BE) epithelium.

ELIGIBILITY:
Inclusion Criteria:

1. Presenting to University of North Carolina (UNC) for routine care upper endoscopy
2. Meet one of the following criteria:

   1. Presenting to UNC for upper endoscopy of GI conditions without esophageal symptomology for with no history of gastroesophageal reflux disease (GERD) or other esophageal condition affecting the epithelium (asymptomatic controls), OR,
   2. History of dysplastic or non-dysplastic Barrett's Esophagus with prague criteria C1+ or M3+
3. Aged 18 to 80
4. Able to read, comprehend, and understand the informed consent document.

Exclusion Criteria:

1. Prior esophageal surgery (uncomplicated nissen fundoplication OK)
2. Pregnant women
3. Unable to provide written informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Wax, Ph.D., Principal Investigator — Professor
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- OCT of Esophagus: All participants who were able to swallow the OCT probe had optical coherence tomography (OCT) imaging of the esophagus, with measurements in at least 5 locations.
Period: Overall Study
Arm/Group | OCT of Esophagus
Started | 53
Completed | 37
Not Completed | 16
Not completed — unable to swallow OCT probe | 16

BASELINE CHARACTERISTICS:
Arm/Group | OCT of Esophagus
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 53
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 53
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 53
Stage of Barrett's Esophagus [Count of Participants; unit: Participants]
  non-dysplastic Barrett's Esophagus | 8
  Barrett's Esophagus with low grade dysplasia | 24
  Barrett's Esophagus with high grade dysplasia | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Imaged Sites Correctly Categorized as Squamous Mucosa
Description: Percentage of imaged sites correctly categorized by OCT as squamous mucosa when compared to endoscopy.
Time Frame: at baseline
Population: Participants who completed the study.
Measure: Number; unit: percentage of imaged sites
Arm/Group | OCT of Esophagus
Number analyzed (Participants) | 37
percentage of imaged sites | 93.1

2. Primary Outcome: Percentage of Imaged Sites Correctly Categorized as Barrett's Mucosa
Description: Percentage of images site correctly categorized by OCT as Barrett's mucosa when compared to endoscopy.
Time Frame: at baseline
Population: Participants who completed the study.
Measure: Number; unit: percentage of imaged sites
Arm/Group | OCT of Esophagus
Number analyzed (Participants) | 37
percentage of imaged sites | 84.6

3. Secondary Outcome: Percentage of Imaged Sites With Adequate Tissue Contact to Acquire a High Quality Image
Description: Percentage of imaged sites that achieved adequate tissue contact to acquire high quality OCT images.
Time Frame: at baseline
Population: Participants who completed the study.
Measure: Number; unit: percentage of imaged sites
Arm/Group | OCT of Esophagus
Number analyzed (Participants) | 37
percentage of imaged sites | 80.5

ADVERSE EVENTS:
Time Frame: 1 week
Description: Subjects were contacted 1 week after OCT imaging to assess any adverse events.
Arm/Group | OCT of Esophagus
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 8/53
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OCT of Esophagus (N=53)
sore throat (Surgical and medical procedures) | 4
bloating (Surgical and medical procedures) | 1
nausea / vomiting (Surgical and medical procedures) | 1
epigastric pain (Surgical and medical procedures) | 1
esophageal pain (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT03434834/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/34/NCT03434834/Prot_SAP_001.pdf